CLINICAL TRIAL: NCT01440569
Title: A Phase 3b, Open-Label, Single Arm Study to Evaluate the Safety and Efficacy of Cobicistat-boosted Darunavir Plus Two Fully Active Nucleoside Reverse Transcriptase Inhibitors in HIV-1 Infected, Antiretroviral Treatment-Naïve and -Experienced Adults With No Darunavir Resistance-associated Mutations
Brief Title: Safety and Efficacy of Cobicistat-boosted Darunavir in HIV Infected Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-216-0130; 2011-003501-22 (EudraCT Number)
Record Dates: First submitted 2011-09-22; First posted 2011-09-26 (Estimated); Results first posted 2014-10-28 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-10

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: HIV-1; HIV; Treatment Naïve; Treatment Experienced
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Cobicistat; Darunavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- COBI-boosted DRV (Experimental): Participants will receive DRV+COBI+2 investigator-selected NRTIs for 48 weeks, and may continue their regimen in the open-label rollover phase.
  Interventions: Drug: COBI; Drug: DRV; Drug: NRTIs

INTERVENTIONS:
Drug: COBI — 150 mg tablet administered orally with food once daily
  Other Names: Tybost®; GS-9350
Drug: DRV — 800 mg (2 x 400 mg tablets) administered orally with food once daily
  Other Names: Prezista®; TMC114
Drug: NRTIs — Participants will receive 2 nucleoside analogue reverse transcriptase inhibitors (NRTIs) selected by the investigator after resistance testing at screening and administered according to prescribing information. NRTIs may include emtricitabine (FTC)/tenofovir disoproxil fumarate (TDF), zidovudine+FTC/TDF, abacavir (ABC)+TDF, ABC+FTC/TDF, ABC+lamivudine (3TC), or didanosine (DDI)+FTC.

SUMMARY:
This study is to evaluate the safety and tolerability of cobicistat-boosted darunavir plus two fully active nucleoside analogue reverse transcriptase inhibitors in HIV 1 infected, antiretroviral treatment-naive and treatment-experienced adults with no darunavir (DRV) resistance-associated mutations.

After the Week 48 Visit, participants will be given the option to participate in an open-label rollover phase to receive cobicistat and attend visits every 12 weeks until it becomes commercially available, or until Gilead Sciences elects to terminate development of cobicistat.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years males or non-pregnant females
* Ability to understand and sign a written informed consent form
* General medical condition that does not interfere with the assessments and the completion of the trial
* Treatment Naive: No prior use of any approved or investigational antiretroviral drug for any length of time OR
* Treatment Experienced: Stable antiretroviral regimen for at least 12 weeks prior to screening
* Plasma HIV-1 RNA levels ≥ 1000 copies/mL at Screening
* Screening genotype report shows full sensitivity to two nucleoside analogue reverse transcriptase inhibitors (NRTIs) and no darunavir resistance-associated mutations
* Normal electrocardiogram (ECG)
* Hepatic transaminases ≤ 2.5 × upper limit of normal (ULN)
* Total bilirubin ≤ 1.5 mg/dL
* Adequate hematologic function
* Serum amylase ≤ 2 × ULN and serum lipase ≤ 3 × ULN
* Adequate renal function: Estimated glomerular filtration rate ≥ 80 mL/min
* Females of childbearing potential must agree to utilize protocol-recommended methods of contraception, or be nonheterosexually active, practice sexual abstinence or have a vasectomized partner from Screening throughout the duration of the study period and for 30 days following the last dose of study drug.
* Male subjects must agree to utilize protocol-recommended methods of contraception during heterosexual intercourse from the Screening visit, throughout the duration of the study and for 30 days following discontinuation of investigational medicinal product or be nonheterosexually active, practice sexual abstinence, or be vasectomized.

Exclusion Criteria:

* Previous or current use of darunavir
* A new AIDS-defining condition diagnosed within the 30 days prior to Screening
* Females who are breastfeeding
* Positive serum pregnancy test (if female of childbearing potential)
* Proven or suspected acute hepatitis in the 30 days prior to study entry
* Subjects receiving drug treatment for hepatitis C virus (HCV), or subjects who are anticipated to receive treatment for HCV during the course of the study
* Have a history of ongoing active liver disease or experiencing decompensated cirrhosis irrespective of liver enzyme levels
* Have an implanted defibrillator or pacemaker
* Current alcohol or substance use that may interfere with subject study compliance
* A history of malignancy within the past 5 years or ongoing malignancy other than cutaneous Kaposi's sarcoma
* Active, serious infections requiring parenteral antibiotic or antifungal therapy within 30 days prior to Baseline
* Participation in any other clinical trial
* Any other clinical condition or prior therapy that would make the subject unsuitable for the study or unable to comply with the dosing requirements.
* Subjects receiving ongoing therapy with any of the medications, including drugs not to be used with cobicistat, darunavir, or investigator selected NRTIs; or subjects with any known allergies to cobicistat tablets, darunavir tablets or contraindications for the 2 NRTIs as part of the regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marshall Fordyce, MD, Study Director — Gilead Sciences
Locations (49):
- United States (48):
  - Spectrum Medical Group, Phoenix, Arizona
  - Long Beach Education and Research Consultants, PC, Long Beach, California
  - Peter J Ruane MD Inc., Los Angeles, California
  - Anthony Mills MD Inc, Los Angeles, California
  - Stanford University, Palo Alto, California
  - Kaiser Permanente Medical Group, Sacramento, California
  - La Playa Medical Group and Clinical Research, San Diego, California
  - Metropolis Medical, San Francisco, California
  - Apex Research LLC, Denver, Colorado
  - Dupont Circle Physician's Group, Washington D.C., District of Columbia
  - Whitman-Walker Health, Washington D.C., District of Columbia
  - Gary J. Richmond,M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Wohlfeiler, Piperato and Associates, LLC, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - St. Joseph's Comprehensive Research Institute, Tampa, Florida
  - Atlanta ID group, Atlanta, Georgia
  - Infectious Disease Specialists of Atlanta, Decatur, Georgia
  - Mercer University, Macon, Georgia
  - Hawaii Center for AIDS, University of Hawaii, Honolulu, Hawaii
  - Howard Brown Health Center, Chicago, Illinois
  - Northstar Medical Center, Chicago, Illinois
  - Johns Hopkins University, Lutherville, Maryland
  - Community Research Initiative of New England, Boston, Massachusetts
  - Be Well Medical Center, Berkley, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Central West Clinical Research Inc, Saint Louis, Michigan
  - HIV Program Hennepin County Medical Center, Minneapolis, Minnesota
  - Saint Michael's Medical Center, Newark, New Jersey
  - South Jersey Infectious Disease, Somers Point, New Jersey
  - North Shore University Hospital / Division of Infectious Diseases, Manhasset, New York
  - Greiger Clinic, Mount Vernon, New York
  - Beth Israel Medical Center, New York, New York
  - Carolinas Medical Center-Myer's Park Infectious Disease Clinic, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Health Services, Winston-Salem, North Carolina
  - University of PA, Philadelphia, Pennsylvania
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
  - Central Texas Clinical Research, Austin, Texas
  - Trinity Health and Wellness Center/AIDS Arms, Inc., Dallas, Texas
  - Southwest Infectious Disease Clinical Research, Inc., Dallas, Texas
  - Tarrant County Infectious Disease, Fort Worth, Texas
  - Therapeutic Concepts, PA, Houston, Texas
  - Gordon Crofoot MD, PA, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research & Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
  - Swedish Medical Center, Seattle, Washington
- Clinical Research Puerto Rico, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at a total of 56 study sites in the United States. The first participant was screened on 22 September 2011. The last study visit occurred on 30 October 2015.
Pre-assignment Details: 397 participants were screened.
Groups:
- Treatment-Naive: Treatment-naive participants received darunavir (DRV; 800 mg; 2 × 400 mg tablets) + cobicistat (COBI; 1 × 150 mg tablet) once daily + two nucleoside analogue reverse transcriptase inhibitors (NRTIs; per prescribing information) for 48 weeks, and may have continued their regimen in the open-label rollover phase.
- Treatment-Experienced: Treatment-experienced participants received DRV (800 mg; 2 × 400 mg tablets) + COBI (1 × 150 mg tablet) once daily + two NRTIs (per prescribing information) for 48 weeks, and may have continued their regimen in the open-label rollover phase.
Period: Main Study
Arm/Group | Treatment-Naive | Treatment-Experienced
Started | 296 | 18
Enrolled and Treated | 295 | 18
Completed | 260 | 14
Not Completed | 36 | 4
Not completed — Enrolled but not treated | 1 | 0
Not completed — Adverse Event | 9 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Investigator's Discretion | 1 | 1
Not completed — Withdrew Consent | 7 | 1
Not completed — Lost to Follow-up | 13 | 2
Not completed — Subject Non-Compliance | 3 | 0
Not completed — Protocol Violation | 1 | 0
Period: Open-Label Rollover Phase
Arm/Group | Treatment-Naive | Treatment-Experienced
Started | 251 (9 participants who completed the Main Study did not enroll into the Rollover Phase.) | 13 (1 participant who completed the Main Study did not enroll into the Rollover Phase.)
Completed | 204 | 7
Not Completed | 47 | 6
Not completed — Adverse Event | 3 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Lack of Efficacy | 2 | 0
Not completed — Investigator's Discretion | 3 | 1
Not completed — Withdrew Consent | 11 | 1
Not completed — Lost to Follow-up | 26 | 3
Not completed — Subject Non-Compliance | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: participants who were enrolled into the study and received at least one dose of study drug.
Groups:
- Treatment-Naive: Treatment-naive participants received DRV (800 mg; 2 × 400 mg tablets) + COBI (1 × 150 mg tablet) once daily + two NRTIs (per prescribing information) for 48 weeks, and may have continued their regimen in the open-label rollover phase.
- Total: Total of all reporting groups
Arm/Group | Treatment-Naive | Treatment-Experienced | Total
Number analyzed (Participants) | 295 | 18 | 313
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10.3) | 45 (10.9) | 36 (10.6)
Gender [Count of Participants; unit: Participants]
  Female | 29 | 5 | 34
  Male | 266 | 13 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 4 | 68
  Not Hispanic or Latino | 231 | 14 | 245
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  White | 176 | 11 | 187
  Black or African Heritage | 101 | 7 | 108
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 4 | 0 | 4
  Native Hawaiian or Pacific Islander | 2 | 0 | 2
  Other | 8 | 0 | 8
CD4 Count (cells/mm^3) [Mean (Standard Deviation); unit: cells/mm^3] | 378.2 (199.94) | 197.8 (214.30) | 367.8 (204.79)
HIV-1 RNA (log10 copies/mL) [Mean (Standard Deviation); unit: log10 copies/mL] | 4.8 (0.76) | 4.8 (1.04) | 4.8 (0.78)
Background Antiretroviral Regimen [Number; unit: participants] — 3TC, lamivudine (Epivir®); ABC, abacavir; ABC/3TC, abacavir/lamivudine coformulation; AZT, azidothymidine or zidovudine; DDI, didanosine; FTC, emtricitabine (Emtriva®); FTC/TDF, emtricitabine/tenofovir disoproxil fumarate coformulation (Truvada®); TDF, tenofovir disoproxil fumarate (Viread®)
  participants
    FTC/TDF | 291 | 10 | 301
    AZT+FTC/TDF | 0 | 5 | 5
    ABC+TDF | 2 | 1 | 3
    ABC+FTC/TDF | 1 | 1 | 2
    ABC/3TC | 1 | 0 | 1
    DDI+FTC | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Onset of Any Treatment-emergent Grade 3 or 4 Adverse Event Between Baseline and Week 24
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
percentage of participants | 5.4 | 11.1

2. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA < 50 Copies/mL at Week 24 (Snapshot Analysis)
Time Frame: Week 24
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
percentage of participants | 83.7 | 61.1

3. Secondary Outcome: Percentage of Participants Achieving HIV-1 RNA < 50 Copies/mL at Week 48 (Snapshot Analysis)
Time Frame: Week 48
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
percentage of participants | 82.7 | 50.0

4. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 24
Time Frame: Baseline; Week 24
Population: Full Analysis Set; the Missing = Excluded method was used, where participants with missing data were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
cells/μL | 145 (131.6) | 99 (161.9)

5. Secondary Outcome: Change From Baseline in CD4+ Cell Count at Week 48
Time Frame: Baseline; Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
cells/µL | 194 (152.1) | 121 (157.0)

6. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-emergent Adverse Event and Any Treatment-emergent Adverse Event Leading to Discontinuation of Study Drug Through Week 24
Time Frame: Up to 24 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
percentage of participants
  Any treatment-emergent adverse event (TEAE) | 88.1 | 83.3
  Any TEAE that led to study drug discontinuation | 5.1 | 0

7. Secondary Outcome: Percentage of Participants Experiencing Any Treatment-emergent Adverse Event and Any Treatment-emergent Adverse Event Leading to Discontinuation of Study Drug Through Week 48
Time Frame: Up to 48 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Treatment-Naive | Treatment-Experienced
Number analyzed (Participants) | 295 | 18
percentage of participants
  Any treatment-emergent adverse event (TEAE) | 91.5 | 88.9
  Any TEAE that led to study drug discontinuation | 5.4 | 0

ADVERSE EVENTS:
Time Frame: Up to a maximum of 204.4 weeks (average: 139.2 weeks)
Description: Safety Analysis Set
Arm/Group | Treatment-Naive | Treatment-Experienced
Serious Adverse Events (participants affected / at risk) | 45/295 | 5/18
Other Adverse Events (participants affected / at risk) | 261/295 | 16/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive (N=295) | Treatment-Experienced (N=18)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 1
Furuncle (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Drug dependence (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 2 | 0
Suicide attempt (Psychiatric disorders) | 4 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-Naive (N=295) | Treatment-Experienced (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 10 | 1
Abdominal pain (Gastrointestinal disorders) | 23 | 1
Abdominal pain lower (Gastrointestinal disorders) | 4 | 1
Abdominal pain upper (Gastrointestinal disorders) | 13 | 1
Constipation (Gastrointestinal disorders) | 13 | 1
Diarrhoea (Gastrointestinal disorders) | 99 | 8
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 18 | 1
Haemorrhoids (Gastrointestinal disorders) | 22 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 80 | 3
Tongue pigmentation (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 9 | 1
Vomiting (Gastrointestinal disorders) | 34 | 3
Chest pain (General disorders) | 12 | 1
Fatigue (General disorders) | 35 | 0
Pyrexia (General disorders) | 21 | 3
Seasonal allergy (Immune system disorders) | 15 | 0
Acarodermatitis (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 33 | 1
Conjunctivitis (Infections and infestations) | 16 | 0
Folliculitis (Infections and infestations) | 16 | 0
Gastroenteritis viral (Infections and infestations) | 6 | 1
Herpes zoster (Infections and infestations) | 7 | 1
Influenza (Infections and infestations) | 20 | 2
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 37 | 4
Onychomycosis (Infections and infestations) | 7 | 1
Pharyngitis (Infections and infestations) | 24 | 0
Rash pustular (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 33 | 4
Syphilis (Infections and infestations) | 25 | 0
Tooth abscess (Infections and infestations) | 10 | 2
Upper respiratory tract infection (Infections and infestations) | 70 | 2
Vaginal infection (Infections and infestations) | 1 | 1
Vulvovaginitis (Infections and infestations) | 0 | 1
Vulvovaginitis trichomonal (Infections and infestations) | 1 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 4 | 1
Contusion (Injury, poisoning and procedural complications) | 7 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 5 | 1
Weight decreased (Investigations) | 4 | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 10 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 20 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Penile wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Squamous cell carcinoma of the vulva (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Amnesia (Nervous system disorders) | 3 | 1
Cerebral atrophy (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 50 | 3
Post herpetic neuralgia (Nervous system disorders) | 1 | 1
Abnormal dreams (Psychiatric disorders) | 12 | 1
Alcohol abuse (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 19 | 3
Depression (Psychiatric disorders) | 37 | 0
Drug dependence (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 18 | 1
Dysuria (Renal and urinary disorders) | 6 | 1
Proteinuria (Renal and urinary disorders) | 3 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 8 | 1
Uterine malposition (Reproductive system and breast disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 27 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 17 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 12 | 2
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 1
Rash (Skin and subcutaneous tissue disorders) | 39 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 2 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 2
Tooth extraction (Surgical and medical procedures) | 1 | 1
Hypertension (Vascular disorders) | 17 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years